CLINICAL TRIAL: NCT05014945
Title: Effect of Combination Therapy With Atelocollagen in Epidural Nerve Block in Patients With Chronic Low Back Pain From Degenerative Lumbar Spine: Pilot Study
Brief Title: Combination Therapy With Atelocollagen in Epidural Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Ji Yeong Kim, Associate Professor, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-2021-0180
Record Dates: First submitted 2021-07-22; First posted 2021-08-20 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Degenerative Lumbar Spine Disease

STUDY DESIGN:
Intervention Model Description: Patients with chronic low back pain due to degenerative spinal disease for more than 6 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atelocollagen group (Experimental): After obtaining informed consent for the study, epidural nerve block was performed. The patient is asked to return to the outpatient clinic of the pain center after 2 weeks. At this time, when the NRS of back pain does not improve by more than 50% compared to before the epidural nerve block and the cross-sectional area of the multifidus muscle using ultrasound is 5 cm2 or less, final enrollment is decided. The evaluation of the cross-sectional area and thickness of the multifidus muscle using ultrasound is performed with the patient prone, and the cross-sectional area of the multifidus muscle is measured at the same position as the level of the lesion on MRI.
  Interventions: Procedure: (atelocollagen group)

INTERVENTIONS:
Procedure: (atelocollagen group) — Epidural nerve block and atelocollagen injection into the multifidus muscle were performed sequentially. The target level is determined by the clinician by combining the pre-MRI and the patient's symptoms. All procedures are performed under the guidance of fluroscopy. For epidural nerve block, use 10cc of 0.9% normal saline mixed with 3000IU of hyaluronidase to be injected. After the epidural nerve block, a solution of 1 mL of atelocollagen mixed with 1 mL of 1% lidocaine is injected into the multifidus muscle to complete the entire procedure.

SUMMARY:
"In this study, the investigators plan to evaluate muscle mass and pain relief 4 weeks after performing epidural nerve block and Type I porcine atelocollagen injection into multifidus muscle in patients with chronic low back pain due to degenerative spinal disease for more than 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for epidural nerve block for lower back pain
2. Patients over 21 years of age
3. Back pain lasting more than 6 months
4. Patients with ineffective or insignificant effects of conventional drugs and nerve block for back pain
5. Patients with spinal stenosis or disc herniation at the lumbar 4-5 or lumbar 5-sacral 1 level on MRI, and the cross-sectional area of the multifidus muscle at the lesion site is less than 5 cm2 when measured by ultrasound.

Exclusion Criteria:

1. When the degree of low back pain is 3 points or less on the 11-scale numeric rating scale (hereafter NRS)
2. If lower back pain has rapidly worsened within the last week
3. If you have other diseases that may cause low back pain: osteoarthritis of the hip joint, cancer, inflammatory arthritis, spondylitis, fibromyalgia, complex regional pain syndrome, herpes zoster, postherpetic neuralgia, etc.
4. When a diagnostic epidural nerve block is planned
5. In the case of receiving conservative treatment, procedure, or surgery other than oral drugs such as epidural nerve block or proliferation treatment for the treatment of lower back pain within 4 weeks of screening
6. When the low back pain assessed by NRS decreased by more than 50% after epidural nerve block in screening
7. If back surgery is planned within 3 months of the procedure
8. When NRS and ODI measurements cannot be made
9. When collagen injection is contraindicated (eg when allergic to swine)
10. Pregnant women
11. If you cannot read or agree to the consent form
12. If you are unable to sign the consent form yourself

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
cross-sectional area of the multifidus muscle | 28 days after atelocollagen injection
  Changes in the cross-sectional area of the multifidus muscle at the 4th week of the intervention compared to before the intervention (measured value using ultrasound at outpatient).

SECONDARY OUTCOMES:
numeric rating score | 28 days after atelocollagen injection
  numeric rating score, Score range from 0 to 100. Higher scores mean a worst outcome.
oswestry disability index | 28 days after atelocollagen injection
  oswestry disability index, Score range from 0 to 50. Higher scores mean a worst outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Ji Yeong Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No